CLINICAL TRIAL: NCT06373471
Title: Improving Quality of Life in Older Patients With Frailty and Hematological Cancer Through Geriatric Assessment and Treatment; A Randomized Controlled Trial. IMPROVE
Brief Title: Improving Quality of Life in Older Patients With Frailty and Hematological Cancer Through Geriatric Assessment
Acronym: IMPROVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Velux Fonden (Other); Danish Cancer Research Foundation (Other); The Dagmar Marshall Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20230101
Record Dates: First submitted 2024-04-04; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Hematologic Malignancy; Treatment Adherence; Treatment Complication; Frailty; Quality of Life
Keywords: Comprehensive Geriatric Assessment
MeSH Terms: conditions — Hematologic Neoplasms; Treatment Adherence and Compliance; Frailty | interventions — Geriatric Assessment; Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Comprehensive Geriatric Assessment and treatment
  Interventions: Other: Comprehensive geriatric assessment (CGA) and treatment
- Control (No Intervention): Standard hematological evaluation of comorbidity and needs during hematological cancer treatment.

INTERVENTIONS:
Other: Comprehensive geriatric assessment (CGA) and treatment — CGA and treatment is as an outpatient evaluation by a geriatric medical specialist and nurse. Specific CGA components in this study include:
  * Assessment of comorbidity and treatments
  * Review of medications including potential adjustment
  * Assessment of current symptoms and health related issues including geriatric syndromes such as depression, dementia, delirium, nutritional problems, falls and fatigue
  * Objective examination including blood tests and electrocardiogram
  * Assessment of activities of daily living (ADL) and instrumental ADL through standardized questionnaires
  * Assessment of domestic conditions, including need for assistance
  * Assessment of physical function Based on findings, the geriatrician will initiate relevant interventions and follow-up as required
  Arms: Intervention arm

SUMMARY:
The Improve study is a randomized controlled trial investigating the efficacy of adding comprehensive geriatric assessment and treatment to standard of care compared with standard of care in older, frail patients with hematological cancer. The investigators aim to recruit 152 study participants who will be randomized 1:1 to intervention- or control group. Study participants in the intervention group will receive the intervention comprehensive geriatric assessment and treatment integrated in the cancer treatment. Study participants in the control group will receive cancer treatment and evaluation of comorbidity and frailty as is usual standard at Department of Hematology. Primary endpoint is elderly functional Index at 12 weeks.

DETAILED DESCRIPTION:
RESEARCH PLAN

STUDY DESIGN IMPROVE aims to investigate the efficacy of adding comprehensive geriatric assessment (CGA) and treatment to standard of care compared with standard of care in older, frail patients with hematological cancer. The investigators aim to recruit 152 study participants who will be randomized 1:1 to intervention- or control group. Study participants in the intervention group will receive the intervention CGA and treatment integrated in the cancer treatment. Study participants in the control group will receive cancer treatment and evaluation as well as management of comorbidity, frailty and needs as is the current standard at Departments of Hematology.

PARTICIPANTS AND TIMELINES One hundred and fifty two patients complying with inclusion and exclusion criteria detailed below will be recruited at participating Hematological Departments in Denmark. Study period is 52 weeks for each study participant.

INTERVENTIONS AND ASSESSMENTS Hematological treatment plan Study participants will be given a hematological cancer treatment plan according to standard guidelines at the discretion of the treating physician at the Department of Hematology. The hematological treatment plan will not be altered because of participation in IMPROVE study. Data on whether the cancer treatment is prescribed with a reduced dose-intensity due to frailty or later reduced due to toxicity will be collected.

CGA and treatment CGA and treatment will be performed before or after initiation of hematological cancer treatment, and within 6 weeks from inclusion. Performing CGA shall not delay initiation of hematological cancer treatment if immediate treatment is necessary. A geriatrician together with a geriatric nurse will perform CGA at the Department of Geriatric Medicine. CGA is more thoroughly described elsewhere in this report. Based on CGA findings, the geriatrician will initiate relevant further investigation(s), intervention(s) and treatment(s) if indicated.

Assessment of functional status The investigators will record the patients exercise habits via a short interview with the patient. The interview contains two questions concerning exercise habits derived from the Survey of Health, Ageing and Retirement in Europe (SHARE). Furthermore objective simple physical muscle strength tests will be applied to assess upper and lower extremity functioning.

Physical tests Physical tests will be assessed at baseline and at 12 and 26 weeks follow-up. Physical tests will be 30 seconds chair stand test (30s-CST) and handgrip strength

Treatment toxicity and adherence to the hematological treatment plan

Data will be collected at the beginning of each treatment cycle until 26 weeks after inclusion. The following data will be collected:

* Treatment type.
* Whether the treatment is a standard regimen, a dose-intensity reduced regimen or a study treatment from another clinical trail.
* Whether the hematological treatment plan has been changed, including reduction of dosage, delay of treatment or preterm end of treatment and the reason for change of treatment plan.
* Treatment toxicity using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCICTCAE v5.0) for selected groups of toxicity
* Date and reason for discontinuation of cancer treatment until treatment completion or 26 weeks after initiation, whichever comes first.

Review of medications Information about polypharmacy (more than 5 daily drugs) will be collected from patients´ personal electronic file of prescriptions and medication purchases at baseline and at 12- and 26-week follow-up.

Hospitalization and survival Patients will be followed through a review of medical records for number and duration of unplanned hospitalizations and overall, and cancer-specific survival at 26- and 52-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years
* New diagnosis or progression/relapse of acute leukemia, chronic myeloid leukemia, chronic lymphocytic leukemia, myelodysplastic syndrome, lymphoma, multiple myeloma, chronic myelomonocytic leukemia or myelofibrosis
* Scheduled systemic cancer treatment or initiated systemic cancer treatment within 6 weeks
* Geriatric 8 frailty score of ≤14 at screening
* Life expectancy > 6 months
* Not hospitalized at the time of inclusion

Exclusion Criteria:

* Current systemic treatment for other coexisting cancer. Patients receiving anti-hormone treatment for breast cancer or prostate cancer are not excluded, if no evidence of disease progression (radiological/biochemical) in past 3 months or if treatment is adjuvant.
* Having consulted a geriatric outpatient clinic past 6 months
* Patients in need of specialized neuro-rehabilitation
* Unable to understand Danish
* Unable to give written informed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Elderly functional Index | 12 and 26 weeks after inclusion
  The Elderly Functional Index (ELFI) is calculated using the physical functioning, role functioning, and social functioning of the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) core 30, and the mobility item of the EORTC-QLQ-elderly 14 (ELD14) questionnaire. ELFI is calculated at baseline and at 12- and 26- week follow-up. Maximum value of ELFI is 100. Minimum value of ELFI is 0. Higher score indicates higher function.

SECONDARY OUTCOMES:
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). | 12 and 26 weeks after inclusion
  The questionnaire contains functional and symptom subscales. Maximum value for scales is 100 and minimum values is 0. A higher score indicates higher function for functional scales and more symptoms for symptom scales.
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Elderly14 (EORTC QLQ-Eld14). | 12 and 26 weeks after inclusion
  The questionnaire contains functional scales and symptom scales. Maximum value for scales is 100 and minimum values is 0. A higher score indicates higher function for functional scales and more symptoms for symptom scales
Handgrip strength | 12 and 26 weeks after inclusion
  Handgrip strength is measured in kilograms with a handgrip dynamometer
30-second chair stand test | 12 and 26 weeks after inclusion
  30-second chair stand test is measured in number of stand-up-and-sit-downs in 30 seconds
Treatment toxicity | Baseline, 12 and 26 weeks after inclusion
  Endpoint is assessed as prevalence of grade > 1 adverse events according to Common Terminology Criteria for Adverse Events Version 5.0 at baseline, 12 and 26 weeks after inclusion
Adherence to hematological cancer treatment | 12 and 26 weeks after inclusion
  Alterations to original cancer treatment plan yes/no
Polypharmacy yes/no | 12 and 26 weeks after inclusion
  Polypharmacy is defined as use of 5 or more daily medications
Unplanned hospital admissions | 26 and 52 weeks after inclusion
  rates and hospital days
Overall and cancer specific survival | 26 and 52 weeks after inclusion
  survival proportion and cancer specific survival proportion

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Frederiksen, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No
The IPD sharing plan is to assess the possibility of publishing IPD or part of IPD in a way that is allowed taken GDPR into account.